CLINICAL TRIAL: NCT06262620
Title: The Comparison of Endobronchial Ultrasound-guided Transbronchial Needle Aspiration, Mediastinal Cryobiopsy Via a Tunnel, and Forceps Biopsy Via a Tunnel in Diagnosing Mediastinal Lymphadenopathy: a Multicenter Randomised Controlled Trial.
Brief Title: The Comparison of EBUS-TBNA, TBMC Via a Tunnel, and TBFB Via a Tunnel in Diagnosing Mediastinal Lymphadenopathy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022-NHLHCRF-LX-01-0201-06
Record Dates: First submitted 2024-02-01; First posted 2024-02-16 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Lymphadenopathy Hilar; Lymphadenopathy Mediastinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EBUS-transbronchial needle aspiration (Experimental): Participants would undertake EBUS-transbronchial needle aspiration.
  Interventions: Procedure: EBUS-TBNA
- EBUS-transbronchial mediastinal cryobiopsy via a tunnel (Experimental): Participants would undertake EBUS-transbronchial mediastinal cryobiopsy via a tunnel.
  Interventions: Procedure: EBUS-TBMC via a tunnel
- EBUS-transbronchial forceps biopsy via a tunnel (Experimental): Participants would undertake EBUS-transbronchial forceps biopsy via a tunnel.
  Interventions: Procedure: EBUS-TBFB via a tunnel

INTERVENTIONS:
Procedure: EBUS-TBNA — A 22G biopsy needle was insert into the lesion through tracheal-bronchial wall under real-time EBUS guided by bronchoscopist. Needle punctures were performed by using the jabbing method. Once it is confirmed that the puncture needle is within the target lesion, the puncture needle is moved back and forth while suction (An empty 50 ml syringe was connected to the port at the end of the puncture needle and aspirated to 20 ml maintained for 20 seconds.) is applied. Each lymph node was operated 5 times.
  Other Names: Endobronchial ultrasound-guided transbronchial needle aspiration.
  Arms: EBUS-transbronchial needle aspiration
Procedure: EBUS-TBMC via a tunnel — First a tunnel between airway wall and mediastinal and/or hilar lesion was made by a puncture dilation catheter (BroncTruTM AK-91-55, Bronchus Inc. Hangzhou, China). The 1.1mm cryoprobe (Erbe 20402-401, ERBE, Tübingen, Germany) entered the target lymph node through the tunnel under direct monitoring of EBUS, and the distance between the tip of the cryoprobe and the border of target lymph node was measured using EBUS. After confirming that the distance was >5 mm, the probe was cooled with liquid carbon dioxide for 5-9 seconds. Then retracted with the bronchoscope and the frozen biopsy tissue. Samples were retrieved by thawing in saline and then fixed in formalin. The same lymph node was operated for 3 times.
  Other Names: endobronchial ultrasound-guided transbronchial mediastinal cryobiopsy via a tunnel.
  Arms: EBUS-transbronchial mediastinal cryobiopsy via a tunnel
Procedure: EBUS-TBFB via a tunnel — Firstly, a tunnel to reach the lymph node is established by making use of a puncture dilation catheter, and a 1.5mm biopsy forceps is pushed into the lymph node through the working channel of the ultrasound bronchoscope. After entering the lymph node, the biopsy forceps were opened proximally to the lymph node, the biopsy forceps were advanced, and then the biopsy forceps were closed distally to the lymph node for each specimen. Each lymph node was operated 5 times.
  Other Names: endobronchial ultrasound-guided transbronchial forceps biopsy
  Arms: EBUS-transbronchial forceps biopsy via a tunnel

SUMMARY:
The goal of this prospective, multi-centre, randomised controlled clinical study is to compare the diagnostic yield and safety of the three biopsy techniques (EBUS-TBNA, EBUS-TBMC via a tunnel, and EBUS-TBFB via a tunnel) in mediastinal/hilar lymph node biopsies.

Participants will divided into EBUS-TBNA group, EBUS-TBMC via a tunnel group, and EBUS-TBFB via a tunnel group at a 1:1:1 ratio by using central, computerized random sequence, and then undertake EBUS-TBNA, EBUS-TBMC via a tunnel, or EBUS-TBFB according to the group.

Researchers will compare the diagnostic yield and incidence of adverse events of the three biopsy techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* At least 1 hilar/mediastinal lesion (short axis ≥ 1 cm) requiring diagnostic bronchoscopy procedure;
* Patients who can understand the purpose of the trial, participate voluntarily and sign an informed consent form.

Exclusion Criteria:

* The lesion is a mediastinal cyst or abscess;
* Combined severe cardiopulmonary diseases, coagulation disorders, poor tolerance to anaesthesia, combined psychiatric disorders or severe neurosis and other relevant contraindications to bronchoscopy;
* EBUS assessment reveals that the lesion is rich in blood flow or adjacent to a large vessel, etc. Consider biopsy to be high risk and inappropriate for continuation of biopsy;
* EBUS did not detect lesions in the hilum and/or mediastinum;
* Those who, in the judgement of the investigator, have poor patient compliance and are unable to complete the study as required due to mental disorders, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-02-18 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
Dignostic yield of EBUS-TBNA, EBUS-TBMC via a tunnel, and EBUS-TBFB | 7 days after the biopsy
  The proportion of participants in whom the biopsy led to a definitive diagnosis.
Incidence rate of adverse events | 7 days after the biopsy
  Symptoms and signs
the adequacy of sample acquisition | 7 days after the biopsy
  Samples resulting in a specific diagnosis or samples with the presence of lymphpcytes were considered as adequate.

SECONDARY OUTCOMES:
the adequacy of sample acquisition | 7 days after the biopsy
  Samples resulting in a specific diagnosis or samples with the presence of lymphpcytes were considered as adequate.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Hou, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Deng MM, Yang Z, Zhong C, Zheng Z, Tong R, Zhou G, Li X, Zhao L, Herth FJF, Hou G. Comparison of diagnostic yield and safety of three endobronchial ultrasound-guided transbronchial biopsy techniques in diagnosing patients with mediastinal/hilar lymphadenopathy: a protocol of multicentre randomised trial in China. BMJ Open. 2025 Sep 23;15(9):e096871. doi: 10.1136/bmjopen-2024-096871. PMID 40987727